CLINICAL TRIAL: NCT03525795
Title: A Phase 1 Study of CPI-1205 With Ipilimumab in Patients With Advanced Solid Tumors Followed by a Phase 2 Basket Study of CPI-1205 With Ipilimumab in Selected Tumor Types Previously Treated With PD-1 or PD-L1 Inhibitors
Brief Title: ORIOn-E: A Study Evaluating CPI-1205 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Constellation Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1205-202
Record Dates: First submitted 2018-04-23; First posted 2018-05-16 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Advanced Solid Tumors
Keywords: Phase 1/2; Oncology; EZH2 Inhibitor
MeSH Terms: conditions — Neoplasms | interventions — (R)-N-((4-methoxy-6-methyl-2-oxo-1,2-dihydropyridin-3-yl)methyl)-2-methyl-1-(1-(1-(2,2,2-trifluoroethyl)piperidin-4-yl)ethyl)-1H-indole-3-carboxamide; Ipilimumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CPI-1205 Combination with ipilimumab (Experimental)
  Interventions: Drug: CPI-1205; Drug: ipilimumab

INTERVENTIONS:
Drug: CPI-1205 — Administered orally
Drug: ipilimumab — Administered intravenously

SUMMARY:
This is a Phase 1/2, multi-center, open-label study of CPI-1205 + ipilimumab in patients with histologically or cytologically confirmed advanced solid tumors. This study is designed to determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of CPI-1205 + ipilimumab in patients with advanced solid tumors. Patients in Phase 2 will be treated at the RP2D of CPI-1205 + ipilimumab.

This study was stopped prior to proceeding to Phase 2; no patients were enrolled in Phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Diagnosis and Prior Treatment:
* Phase 1: Patients with histologically or cytologically confirmed locally advanced (unresectable) or metastatic solid tumors and with progressive disease during or after treatment with a PD-1 or PD-L1-inhibitor who meet one of the following criteria:

  1. Relapsed following or progressed through standard therapy
  2. Have a disease for which no standard effective therapy exists (i.e., a therapy that demonstrates a significant increase in survival)
  3. Not a candidate for standard effective therapy NOTE: In men with prostate cancer, baseline testosterone levels must also be ≤50ng/dL (≤ 2.0nM) and surgical or ongoing medical castration must be maintained throughout the duration of the study.
* Phase 2: Patients with histologically or cytologically confirmed diagnosis of one of the following and with progressive disease during or after treatment with a PD-1 or PD-L1-inhibitor:

  1. Cohort A: unresectable or metastatic melanoma
  2. Cohort B: metastatic NSCLC
  3. Cohort C: advanced or metastatic (stage 4) RCC
  4. Cohort D: unresectable or metastatic urothelial carcinoma (urethra, bladder, ureters, or renal pelvis)
* If patient has known brain metastases, must have stable neurologic status following local therapy for at least 4 weeks without the use of steroids or on stable or decreasing dose of ≤10 mg daily prednisone (or equivalent), and must be without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events (AEs).
* Phase 1: patients may have measurable or non-measurable disease; measurable disease via RECIST 1.1 is required for Phase 2 patients
* Recovery from recent surgery, radiotherapy, chemotherapy or any other anti-cancer therapy to baseline or ≤ Grade 1 (other than alopecia); ≤ Grade 2 neuropathy allowed
* Demonstrate adequate organ function
* Ability to swallow and retain oral medications

Exclusion Criteria:

* Carcinomatous meningitis
* Prior treatment with CTLA-4 inhibitor
* Phase 2 Cohort: ocular melanoma
* Experienced an immune-related adverse event (irAE) that led to permanent discontinuation of prior immunotherapy
* History of severe hypersensitivity reaction to treatment with another monoclonal antibody
* History of interstitial lung disease, idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan; NOTE: history of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Known history of human immunodeficiency virus (HIV) (HIV1/2 antibodies)
* Gastrointestinal (GI) disorder that negatively affects absorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Phase 1: Frequency of Dose-limiting toxicities (DLTs) | 1 year
  The RP2D will be selected based on the PK, pharmacodynamics and overall tolerability of the regimen, but will not exceed the MTD.
Phase 2: Objective response rate | 1 year
  The rate of confirmed complete responses (CR) + partial responses (PR) as determined by RECIST 1.1 criteria

SECONDARY OUTCOMES:
Objective response rate | 1 year
  The rate of confirmed iCR + iPR
Clinical Benefit Rate | 3 months
  The rate of CR + PR + stable disease (SD) after 3 months of treatment as determined by RECIST 1.1 criteria and as the rate of iCR + iPR + iSD after 3 months of treatment by iRECIST criteria
Time to response | 1 year
  The time from day (D) 1 of treatment to the date of first response as determined by RECIST 1.1 and iRECIST criteria
Duration of Response | 1 year
  The time from measurement criteria are first met for CR/PR or iCR/iPR (whichever is first recorded) until the date of recurrence or progressive disease as determined by RECIST 1.1 and iRECIST criteria
Duration of treatment | 1 year
  The time from D1 of treatment until the date treatment is discontinued for any reason
Progression free survival | 6 months
  The time from D1 of treatment to the date of progression or death, whichever occurs first with progressive disease as determined by RECIST 1.1 and iRECIST criteria
Adverse Events | 1 year
  AEs will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 4.03 (CTCAE v4.03).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - START Midwest, Grand Rapids, Michigan
  - The University of Texas - MD Anderson Cancer Center, Houston, Texas
  - South Texas Oncology & Hematology, San Antonio, Texas